CLINICAL TRIAL: NCT04050657
Title: A Randomized Clinical Trial Investigating the Effect of Appointment Intervals on Orthodontic Tooth Alignment
Brief Title: Appointment Intervals and Orthodontic Tooth Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS Project ID: 255727
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-11

CONDITIONS: Orthodontic Treatment
Keywords: orthodontic treatment; alignment; rate of tooth movement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-week appointment interval group (Experimental): Orthodontic patients who come to tighten their braces every 2-weeks.
  Interventions: Other: appointment interval
- Eight-week appointment interval group (Other): Orthodontic patients who come to tighten their braces every every 8-weeks.
  Interventions: Other: appointment interval

INTERVENTIONS:
Other: appointment interval — To change the appointment interval for one group and keep the standard interval for the other group by measuring alignment duration, measured as days needed to align the teeth using full-arch fixed appliances

SUMMARY:
The purpose of this study is to investigate rapidity of tooth alignment in a randomised clinical trial of orthodontic patients allocated randomly into two different appointment intervals groups. First group will be reviewed every two weeks to adjust their braces while the second group will be reviewed every 8 weeks.

DETAILED DESCRIPTION:
Orthodontics is a branch of dentistry concerned primarily with the correction of dental crowding or tooth malalignment. The first phase of fixed appliance orthodontic treatment is concerned with tooth alignment and relies upon a rapid and predictable response of the appliance system to the forces applied by the aligning archwire. The appropriate length of time between orthodontic appointments, generally called the 'appointment interval', has been the subject of debate for many years. Doctors all have their own preferences, based either on what they were taught in their orthodontic specialty programs or on community norms. Little evidence has been presented in the orthodontic literature to support these biases. The appointment interval may influence tooth alignment rates and treatment time along with other variables, such as periodontal status. Accelerating orthodontic tooth movement can significantly reduce treatment duration and the risk of side-effects.

ELIGIBILITY:
Inclusion Criteria:

Subjects should:

1. be aged 12-18 years old;
2. present with a crowded lower arch that requires orthodontic tooth alignment with a fixed appliance;
3. be medically fit and healthy (absence of systemic diseases);
4. have normal weight (according to body mass index measurements BMI);
5. have permanent dentition;
6. have lower incisor irregularity of 5-12 mm;
7. not having complete overbite;
8. be either extraction or non-extraction cases;
9. be able to give informed consent.

Exclusion Criteria:

1. Subjects who have received fixed orthodontic treatment before.
2. Subjects who will be participating in any other intervention trials.
3. Subjects with reported nickel allergy.
4. Subjects who have received antibiotic therapy in the previous six months, or who have any history of juvenile periodontal disease.
5. Subjects who have lower incisor extracted tooth.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to completion of alignment. | 4-10 months.
  To measure the time taken to achieve orthodontic tooth alignment using fixed appliances in two groups of patients treated with different appointment intervals

SECONDARY OUTCOMES:
Level of oral biomarkers | 4-10 months.
  In vivo levels of oral biomarkers derived from gingival crevicular fluid in the periodontal ligament and saliva. Biomarkers associated with orthodontic tooth movement and/or periodontitis will be tested, including biomarkers for tissue damage and inflammatory processes, such as Lactate dehydrogenase (LDH) and Aspartate aminotransferase (AST), biomarkers to asses inflammation in orthodontic movement, such as Myeloperoxidase (MPO) , biomarkers for resolution of organic matrix and bone resorption, such as Cathepsin B, biomarkers for periodontal ligament remodelling, such as Matrix Metalloproteinases (MMPs).
Self-reported pain and discomfort. | 4-10 months.
  At each adjustment visit, subjects will be given a prepared discomfort questionnaire to complete over the following week and to be returned at each subsequent visit. This questionnaire records discomfort by means of a 100 mm visual analogue scale (VAS) at 4 hours, 24 hours, 3 days, and 1 week, using the terms 'very comfortable' and 'very uncomfortable' as peripheral weightings (Seymour, 1982). The VAS score is the distance from the left end of the line to the point of the subject's mark, measured to the nearest millimetre.
Periodontal health. | 4-10 months
  Periodontal health will be measured using established Gingival and Plaque indices. The criteria for plaque index as:
  0: No plaque
  1. A film of plaque adheres to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using probe on the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and the gingival margin, which can be seen with the naked eye.
  3. An abundance of soft matter within the gingival pocket and/or the tooth and gingival margin.
  The criteria for gingival index as:
  0: Normal gingiva.
  1. Mild inflammation: slight change in colour, slight oedema, no bleeding on probing.
  2. Moderate inflammation: moderate glazing, redness, oedema, and hypertrophy, bleeding on probing.
  3. Severe inflammation: marked redness and hypertrophic ulceration, tendency to spontaneous bleeding
Rate of tooth movement | 4-10 months
  Rate of tooth alignment will be calculated from serial dental study casts using Little's Irregularity Index, which measures the horizontal linear contact-point displacement of each mandibular incisor from the adjacent tooth and therefore, represents the sum of the five individual displacements (Little, 1975).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Martyn Cobourne, Principal Investigator — King's College London; Dr. Guy Carpenter, Principal Investigator — King's College London
Locations (1):
- Guy's hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Un-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Zenodo (open-access repository).

REFERENCES:
- [Background] Saloom HF, Papageorgiou SN, Carpenter GH, Cobourne MT. Impact of Obesity on Orthodontic Tooth Movement in Adolescents: A Prospective Clinical Cohort Study. J Dent Res. 2017 May;96(5):547-554. doi: 10.1177/0022034516688448. Epub 2017 Jan 23. PMID 28113000
- [Background] Scott P, DiBiase AT, Sherriff M, Cobourne MT. Alignment efficiency of Damon3 self-ligating and conventional orthodontic bracket systems: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2008 Oct;134(4):470.e1-8. doi: 10.1016/j.ajodo.2008.04.018. PMID 18929262